CLINICAL TRIAL: NCT03233074
Title: Constitution of a Biological Cohort Following Bone Marrow Sampling From MDS or AML Patients and Age-matched Healthy Donors (COSMOS)
Brief Title: Constitution of a Biological Cohort Following Bone Marrow Sampling From MDS or AML Patients and Age-matched Healthy Donors
Acronym: COSMOS
Status: Terminated | Type: Observational
Why Stopped: Achievement of scientific objectives
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0701; 2017-A02088-45 (Other: ANSM)
Record Dates: First submitted 2017-07-17; First posted 2017-07-28 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Cardio-vascular Surgery
Keywords: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Bone Marrow; Mesenchymal stromal cell; Healthy donor
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Myeloid Leukemia patients: For diagnosis purpose, bone marrow sampling is performed for acute myeloid leukemia patients. 2 milliliters of this sample will be collected and analysed for the COSMOS study.
  Interventions: Other: Bone marrow analyses
- Healthy donors: Healthy donors are patients undergoing cardio-vascular surgery for their usual support. During this surgery, 2 milliliters of the bone marrow will be collected, and analysed for the COSMOS study.
  Interventions: Other: Bone marrow analyses

INTERVENTIONS:
Other: Bone marrow analyses — This is a non-interventional study for the constitution of a biobank of bone marrows, in order to further investigate in vitro the cellular properties of bone marrow-isolated mesenchymal stromal cells.
  Other Names: Cellular properties of mesenchymal stromal cells

SUMMARY:
It is of clinical significance to better characterize the intrinsic defects harbored by mesenchymal stromal cells (MSC) in Myelodysplastic syndromes (MDS) and acute myeloid leukemia (AML) context, as compared to physiological conditions. Such research initiative aims to dissect the cross-talk between malignant hematopoietic stem cells (HSC) and their bone marrow (BM) partners in crime, further prospecting for innovative stromal-directed strategies for the treatment of Myelodysplastic syndromes (MDS) and acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are a heterogeneous group of clonal malignancies that are characterized by ineffective hematopoiesis, progressive bone marrow failure, cytogenetic and molecular abnormalities, and increased risk for progression to acute myeloid leukemia (AML). It is a well-accepted theory that MDS and AML originate from primary alterations of hematopoietic stem cells (HSC) compartment, which confer a survival advantage to them at the expense of physiological hematopoiesis. More recently, there is growing evidences regarding the contribution of the bone marrow (BM) microenvironment to the pathogenesis of MDS and AML. Of particular interest, several studies have pointed towards a pivotal role of mesenchymal stromal cells (MSC), one of the main components of the BM niche, in the initiation and propagation of myeloid disorders. In this context, it is of clinical significance to better characterize the intrinsic defects harbored by MSC in MDS and AML context, as compared to physiological conditions. Such research initiative aims to dissect the cross-talk between malignant HSC and their BM partners in crime, further prospecting for innovative stromal-directed strategies for the treatment of MDS and AML.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed myelodysplasia or acute myeloid leukemia (study place: ICLN) - Specific to the cases cohort
* Age-matched healthy donors undergoing a cardiovascular surgery - Specific to the control cohort
* Signed written informed consent form
* Patient affiliated to a social security regimen or beneficiary of the same

Exclusion Criteria:

* Medical history of hematological disorders
* Thrombocytopenia, anemia…
* Patient under guardianship or deprived of his liberty or any condition that may affect the patient's ability to understand and sign the informed consent (art. L.1121-6, L.112-7, L.1211-8, L.1211-9)
* Pregnant or breastfeeding women
* Refusing participation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute Myeloid Leukemia patients undergoing a bone marrow sampling for diagnosis purposes, and healthy donors undergoing cardio-vascular surgery for their usual support.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Changes in cellular properties of mesenchymal stromal cells | Day 0
  Changes in cellular properties of mesenchymal stromal cells isolated from bone marrow aspirates by comparing normal cells (i.e. healthy donors) and MDS/AML cells.

SECONDARY OUTCOMES:
Number of differential biomarkers in mesenchymal stromal cells | Day 0
  Number of differential biomarkers expressed by MDS or AML-derived mesenchymal stromal cells

CONTACTS AND LOCATIONS:
Overall Officials: Denis Guyotat, PhD, Principal Investigator — CHU de Saint-Etienne
Locations (2):
- France (2):
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No